CLINICAL TRIAL: NCT06387472
Title: Adaptive Deployment of DermAI to Evaluate Human Factor of Testing
Brief Title: DermAI to Evaluate Human Factor of Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew Hall, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-007636
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DermAI and Patch Allergen Testing (Experimental): Subjects will have two allergen patches on their forearms for 48 hours. After 48 hours, the patches will be removed and a photograph will be taken where the patches were placed. This photograph will undergo interpretation by a medical professional and by the AI algorithm (DermAI) to evaluate for positive allergic reactions.
  Interventions: Device: AI algorithm to evaluate photographs of skin test patch regions; Device: Allergen Patch

INTERVENTIONS:
Device: AI algorithm to evaluate photographs of skin test patch regions — Interpretation of skin test patch regions via artificial intelligence (AI)
  Other Names: DermAI
Device: Allergen Patch — Contains dime-sized disks which have different substance to which a person may be allergic. Two different patches were used due to the number of allergens being tested. Each patch can only hold 10 allergens and 14 allergens were tested in patients.

SUMMARY:
The purpose of this research is to improve how well remote patch allergy testing works and make sure they are easy and practical for people to use from home.

ELIGIBILITY:
Inclusion Criteria:

- Willing and able to provide informed consent.

Exclusion Criteria:

* Has used topical or oral steroids two weeks prior to patch testing.
* Currently taking immunosuppression agents or is immunocompromised due to medical condition.
* No sunburn or rash at site of testing.
* Women who are breastfeeding or pregnant.
* Treatment with ultraviolet (UV) light (including tanning) during the two weeks prior to visit.
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting patch test area from excess moisture due to showering).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DermAI and Patch Allergen Testing
Started | 151
Completed | 147
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 138
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 45
  White | 83
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 151

OUTCOME MEASURES:

1. Primary Outcome: Classification of Test Site Region Reaction
Description: Number of skin patch interpretations using novel AI algorithms analysis to be in concordant with human review interpretation for the classification of regions within the test panel that either were a reaction (reaction grade 1+) or no reaction (grade 0).
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Count of Units; unit: Skin Patch Interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 1410
Skin Patch Interpretations
  Human Review Interpretation-Grade 0 | 1247
  Human Review Interpretation-Grade 1+ | 163
  AI Model Predication-Grade 0 | 1126
  AI Model Predication-Grade 1+ | 284

2. Secondary Outcome: Classification of Test Site Region Using a 5-point Scale Where Skin Patch Interpretations Were a Grade 0
Description: Number of skin patch interpretations using novel AI algorithms analysis to be in concordant with human review interpretation for the classification of the test site region using a 5-point scale: Grades 0 - 4 with higher scores indicating worse outcome.
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Number; unit: percentage of grade 0 interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 1247
percentage of grade 0 interpretations
  Human Review Interpretation-Grade 0 | 100
  AI Model Predication-Grade 0 | 88.3

3. Secondary Outcome: Classification of Test Site Region Using a 5-point Scale Where Skin Patch Interpretations Were a Grade 1
Description: as for outcome 2
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Number; unit: percentage of grade 1 interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 20
percentage of grade 1 interpretations
  Human Review Interpretation-Grade 1 | 100
  AI Model Predication-Grade 1 | 70

4. Secondary Outcome: Classification of Test Site Region Using a 5-point Scale Where Skin Patch Interpretations Were a Grade 2
Description: as for outcome 2
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Number; unit: percentage of grade 2 interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 132
percentage of grade 2 interpretations
  Human Review Interpretation-Grade 2 | 100
  AI Model Predication-Grade 2 | 85.6

5. Secondary Outcome: Classification of Test Site Region Using a 5-point Scale Where Skin Patch Interpretations Were a Grade 3
Description: as for outcome 2
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Number; unit: percentage of grade 3 interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 8
percentage of grade 3 interpretations
  Human Review Interpretations-Grade 3 | 100
  AI Model Predications-Grade 3 | 100

6. Secondary Outcome: Classification of Test Site Region Using a 5-point Scale Where Skin Patch Interpretations Were a Grade 4
Description: as for outcome 2
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Number; unit: percentage of grade 4 interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 3
percentage of grade 4 interpretations
  Human Review Interpretations-Grade 4 | 100
  AI Model Predications-Grade 4 | 100

7. Secondary Outcome: False Positive Rate
Description: Number of false positive AI interpretations
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Count of Units; unit: Skin Patch Interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 1410
Skin Patch Interpretations | 146

8. Secondary Outcome: False Negative Rate
Description: Number of false negative AI interpretations
Time Frame: 1 week
Population: Six participants were not included in the analysis due to being a part of the pilot phase of the study.
Measure: Count of Units; unit: Skin Patch Interpretations
Units Other Than Participants: Skin Patch Interpretations
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 141
Number analyzed (Skin Patch Interpretations) | 1410
Skin Patch Interpretations | 25

9. Secondary Outcome: Early Termination of Testing
Description: Number of early termination of testing
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 151
Participants | 1

10. Secondary Outcome: Participants That Removed Patches Early
Description: Number of participants that removed patches early
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 151
Participants | 1

11. Secondary Outcome: Adverse Events Related to Allergen Exposure
Description: Number of adverse events related to allergen exposure
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | DermAI and Patch Allergen Testing
Number analyzed (Participants) | 151
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 1 week.
Arm/Group | DermAI and Patch Allergen Testing
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT06387472/Prot_SAP_000.pdf